CLINICAL TRIAL: NCT03797443
Title: Phase IB/II Trial of High Dose Ascorbic Acid (AA) + Nanoparticle Paclitaxel Protein Bound + Cisplatin + Gemcitabine (AA NABPLAGEM) in Patients Who Have Had No Prior Therapy for Their Metastatic Pancreatic Cancer
Brief Title: High Dose Ascorbic Acid (AA) + Nanoparticle Paclitaxel Protein Bound + Cisplatin + Gemcitabine (AA NABPLAGEM) in Patients Who Have Metastatic Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Regulatory Review needed
Sponsor: Piedmont Cancer Institute (Other)
Collaborators: Cancer Research UK (Other); Stand Up To Cancer (Other); Lustgarten Foundation (Other); Destroy Pancreatic Cancer (Other); Translational Genomics Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAN-VITC
Record Dates: First submitted 2018-12-05; First posted 2019-01-09 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Metastatic Pancreatic Cancer; Cancer; Pancreatic; Vitamin C; Ascorbic Acid; Paclitaxel Protein Bound; Cisplatin; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Ascorbic Acid; Taxes; Cisplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Ascorbic Acid Paclitaxel Protein Bound Cisplatin Gemcitabine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AA NABPLAGEM (Experimental): Ascorbic Acid Paclitaxel protein-bound cisplatin gemcitabine
  Interventions: Drug: Ascorbic Acid; Drug: nab paclitaxel; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Ascorbic Acid — Four escalating dose levels are planned in order to determine the MTD for Phase II
  The dose level for Phase II patients will be determined following completion of the Phase 1b study based on response from 3-6 patients receiving the designated dose level of ascorbic acid.
  Other Names: Vitamin C
Drug: nab paclitaxel — 30 minute IV infusions on days 1 and 8 repeated every 21 days, followed by Cisplatin
Drug: Cisplatin — 60minute IV infusion on days 1 and 8 repeated every 21 days followed by Gemcitabine
Drug: Gemcitabine — 30 minute IV infusion on days 1 and 8 repeated every 21 days

SUMMARY:
The purpose of this study is to see if a combination of paclitaxel protein bound (also known as nab-paclitaxel), gemcitabine, and cisplatin when given with high dose Ascorbic Acid will be safe and effective in individuals with untreated metastatic pancreatic cancer.

Vitamin C is a nutrient found in food and dietary supplements. It protects cells and also plays a key role in making collagen (which provides strength and structure to skin, bones, tissues and tendons). High-dose vitamin C may be given by intravenous (IV) infusion (through a vein into the bloodstream) or orally (taken by mouth). When taken by intravenous infusion, vitamin C can reach much higher levels in the blood than when the same amount is taken by mouth. Some human studies of high-dose IV vitamin C in patients with cancer have shown improved quality of life, as well as improvements in physical, mental, and emotional functions, symptoms of fatigue, nausea and vomiting, pain, and appetite loss. Intravenous high-dose ascorbic acid has caused very few side effects in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Histologically or cytologically confirmed metastatic pancreatic adenocarcinoma (with measurable disease according to RECIST 1.1)
* Have a performance status of 0 or 1 on the ECOG performance scale.
* Demonstrate adequate organ function as defined below in Table 4, all screening labs should be performed within 21 days of treatment initiation.
* Female participants of childbearing potential should have a negative serum pregnancy test within 72 hours prior to receiving first dose of study medication.
* Female participants of childbearing potential must be willing to use adequate method of contraception (as outlined in section 4.4.2) for the duration of the trial through one month after the last dose of trial treatment.
* Male participants must agree to use adequate contraception (as outlined in section 4.4.2) for the duration of the trial through one month after the last dose of trial treatment. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.

Exclusion Criteria:

* Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatments in the adjuvant setting with gemcitabine and/or 5-FU or gemcitabine administered as a radiation sensitizer are allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
* Palliative surgery and/or radiation treatment less than 4 weeks prior to initiation of study treatment.
* Exposure to any investigational agent within 4 weeks prior to initiation of study treatment.
* Patients who need constant use of finger stick blood glucose monitoring for tight control of their diabetes being that the ascorbic acid causes false low readings of glucose via that technology (Vasudevan and Hirsch 2014) 39
* Any person with a G6PD deficiency
* History of renal oxalate stones (if type of stone is unknown, need to assess urine oxalates level if >60mg/dL, then patient is not eligible for the study)
* Patient is taking acetaminophen at any dose or any medication that contains acetaminophen within 72 hours of first dose of ascorbic acid
* Hypersensitivity to any of the agents proposed for treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* For female participants: Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the pre-screening or screening visit through one month after the last dose of trial treatment.
* For male participants: Is expecting to impregnate a sexual partner within the projected duration of the trial, starting with the pre-screening or screening visit through one month after the last dose of trial treatment.
* Patients with evidence of iron overload, defined as a transferrin saturation > 45 percent AND serum ferritin > 200 ng/mL (males) or >150 ng/mL (females).
* Current, serious, clinically significant cardiac arrhythmias as determined by the investigator, or patient receiving a digitalis derivative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | approx 63 days
  To determine the maximum tolerated dose (MTD) of high dose ascorbic acid (AA) with triple therapy of nanoparticle paclitaxel protein bound+ cisplatin + gemcitabine (NABPLAGEM) in patients with advanced stage IV metastatic pancreatic cancer
Disease control rate (CR+PR+SD x18 weeks) | approx 63 days
  To determine the preliminary efficacy (Disease control rate of CR+ PR+SD X 18 weeks) of the combination of high dose ascorbic acid (AA) at MTD with triple therapy of nanoparticle albumin- bound paclitaxel + cisplatin + gemcitabine (NABPLAGEM) in patients with advanced stage IV metastatic pancreatic cancer.

SECONDARY OUTCOMES:
Incidence of Treatment | 63 days
  Lab testing will be completed to evaluate standard of care labs for subject safety
Percent of patients who normalize their CA19-9 | 63 days
  Lab testing will be completed to evaluate normalization of CA19-19
Overall survival (OS) | 12 weeks
  Telephone followup will be conducted every 12 weeks from the last dose of treatment to determine survival status
Progression free | approximately 12 weeks from last study treatment ]
  Telephone followup will be conducted every 12 weeks from the last dose of treatment to determine status of disease progression
Changes in patient's self-reported quality of life | 63 days
  Changes in patient's self-reported quality of life will be determined by administering the MD Anderson Symptom Inventory for Gastrointestinal Cancer (MDASI-GI) to assess the severity of multiple gastrointestinal cancer-related syymptoms and the impact of these symptoms of daily functiong.
Changes in patient's self-reported pain levels | 63 days
  Changes in patient's self-reported pain levels will be determined by administering the Brief Pain Inventory (BPI) to assess the severity of pain and the impact of pain on daily functions.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Piedmont Cancer Institute, Fayetteville, Georgia
  - Piedmont Cancer Institute, Newnan, Georgia

IPD SHARING:
Plan to Share IPD: No